CLINICAL TRIAL: NCT03441503
Title: Child HCAHPS: Day of Discharge Survey on an Electronic Interactive Patient Care System
Brief Title: Child HCAHPS: Automated Day of Discharge Survey
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: We were not able to enroll partner hospitals.
Sponsor: Boston Children's Hospital (Other)
Collaborators: GetWellNetwork (Other); Dayton Children's Hospital (Other)
Responsible Party: Principal Investigator, Sara Toomey, Principal Investigator and Director, Center of Excellence for Pediatric Quality Measurement; Chief Experience Officer, Boston Children's Hospital; Assistant Professor of Pediatrics, Harvard Medical School, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: P00001745; U18HS025299 (AHRQ)
Record Dates: First submitted 2018-02-15; First posted 2018-02-22 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Inpatient Experience Survey Administration; Inpatient Experience Survey Response

STUDY DESIGN:
Intervention Model Description: This study is a rapid cycle randomized control trial. Participating units will alternate between the intervention arm (day of discharge survey via inpatient television) and control arm (post-discharge mailed survey). Patients will be assigned to the intervention or control arm depending on the status of their discharging unit. Units will alternate arms throughout the study period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Child HCAHPS: Automated Administration (Experimental): Child HCAHPS: Automated day-of-discharge survey
  On the day of discharge at the hospital, parents will be contacted to solicit survey responses using patient televisions (GetWell) as follows:
  Day 0 (Day of likely discharge): Respondent will be promoted to complete Child HCAHPS on their television as part of the routine discharge process. Respondent will also be asked for their email address to complete post-discharge items and their appropriate contact information will be collected.
  Days 2-42: Standard hospital protocol (i.e., mail, email, or IVR) with the post-discharge questions.
  Interventions: Other: Child HCAHPS: Automated day-of-discharge survey
- Standard Administration of Child HCAHPS (No Intervention): Parents will be contacted to complete Child HCAHPS using the standard protocol for mail, email, or IVR survey administration. The surveys will be administered by the survey vendor contracted by the participating site to administer Child HCAHPS.

INTERVENTIONS:
Other: Child HCAHPS: Automated day-of-discharge survey — Child HCAHPS surveys will be administered on the day of discharge via an electronic interactive patient care system on inpatient televisions.
  Arms: Child HCAHPS: Automated Administration

SUMMARY:
The goal of this study is to identify effective ways to assess the patient and family experience. Specifically, the study will examine automated administration of the Child Hospital Consumer Assessment of Healthcare Providers and Systems (HCAHPS) Survey on the day of discharge through an electronic interactive patient care system. The will be a multisite study that will take place at Boston Children's Hospital (BCH) as well as at several other hospitals across the United States.

DETAILED DESCRIPTION:
Preliminary research conducted by BCH on alternative administration methods of Child HCAHPS has proven promising. Specifically, a pilot of administration on the day of discharge using tablet computers increased response rates, especially among hard to reach groups.

To further explore modes of Child HCAHPS day of discharge administration, the Center of Excellence for Pediatric Quality Measurement (CEPQM) at BCH is collaborating with GetWellNetwork (GetWell), a company that provides interactive education material for patient televisions, to enable parents and guardians to complete Child HCAHPS on the day of discharge from the inpatient television. For this multisite study, parents of hospitalized children from BCH and participating sites will be randomized at the time of discharge to either receiving Child HCAHPS on the day of discharge on the inpatient television or standard Child HCAHPS administration via mail or email. The study will continue for up to six months at each participating site.

ELIGIBILITY:
Inclusion Criteria:

* Their child's hospitalization includes at least one overnight stay

Exclusion Criteria:

* Their child is aged 18 or older during the hospitalization
* Their child is hospitalized with a primary psychiatric diagnosis
* Their child dies during hospitalization
* Their child is in the hospital as a court/law enforcement patient
* Their child is a ward of the state
* Their child was admitted under DCF jurisdiction
* They are not fluent in English or Spanish

Max Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 23578 (Actual)
Dates: Start 2018-04-10 (Actual); Primary Completion 2022-04-10 (Actual); Study Completion 2022-04-10 (Actual)

PRIMARY OUTCOMES:
Child HCAHPS Response Rate | up to 1 year
  Change in response rate to the Child HCAHPS survey

SECONDARY OUTCOMES:
Child HCAHPS Measure Top-Box Scores | up to 1 year
  Change in Child HCAHPS top-box scores (i.e., percent of respondents selecting the most positive response option [0-100%]). Higher top-box scores imply better patient/family experience.
Patient and respondent characteristics | up to 1 year
  Difference in patient/respondent characteristics

CONTACTS AND LOCATIONS:
Overall Officials: Sara Toomey, MD, MPH, MPhil, MSc, Principal Investigator — Boston Children's Hospital, Harvard Medical School
Locations (2):
- United States (2):
  - Boston Children's Hospital, Boston, Massachusetts
  - Dayton Children's Hospital, Dayton, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Toomey SL, Zaslavsky AM, Elliott MN, Gallagher PM, Fowler FJ Jr, Klein DJ, Shulman S, Ratner J, McGovern C, LeBlanc JL, Schuster MA. The Development of a Pediatric Inpatient Experience of Care Measure: Child HCAHPS. Pediatrics. 2015 Aug;136(2):360-9. doi: 10.1542/peds.2015-0966. Epub 2015 Jul 20. PMID 26195542
- [Background] Toomey SL, Elliott MN, Zaslavsky AM, Klein DJ, Ndon S, Hardy S, Wu M, Schuster MA. Variation in Family Experience of Pediatric Inpatient Care As Measured by Child HCAHPS. Pediatrics. 2017 Apr;139(4):e20163372. doi: 10.1542/peds.2016-3372. Epub 2017 Mar 22. PMID 28330970
- [Background] Gurland B, Alves-Ferreira PC, Sobol T, Kiran RP. Using technology to improve data capture and integration of patient-reported outcomes into clinical care: pilot results in a busy colorectal unit. Dis Colon Rectum. 2010 Aug;53(8):1168-75. doi: 10.1007/DCR.0b013e3181d87468. PMID 20628281
- [Background] Martin P, Brown MC, Espin-Garcia O, Cuffe S, Pringle D, Mahler M, Villeneuve J, Niu C, Charow R, Lam C, Shani RM, Hon H, Otsuka M, Xu W, Alibhai S, Jenkinson J, Liu G. Patient preference: a comparison of electronic patient-completed questionnaires with paper among cancer patients. Eur J Cancer Care (Engl). 2016 Mar;25(2):334-41. doi: 10.1111/ecc.12318. Epub 2015 Apr 20. PMID 25899560
- [Background] Turney BW, Reynard JM. Obtaining patient feedback in an outpatient lithotripsy service is facilitated by use of a touch-screen tablet (iPad) survey. Urolithiasis. 2014 Aug;42(4):317-21. doi: 10.1007/s00240-014-0662-3. Epub 2014 Apr 19. PMID 24747981
- [Background] Hofmann JN, Checkoway H, Borges O, Servin F, Fenske RA, Keifer MC. Development of a computer-based survey instrument for organophosphate and N-methyl-carbamate exposure assessment among agricultural pesticide handlers. Ann Occup Hyg. 2010 Aug;54(6):640-50. doi: 10.1093/annhyg/meq038. Epub 2010 Apr 22. PMID 20413416
- [Background] Mullen KH, Berry DL, Zierler BK. Computerized symptom and quality-of-life assessment for patients with cancer part II: acceptability and usability. Oncol Nurs Forum. 2004 Sep 17;31(5):E84-9. doi: 10.1188/04.ONF.E84-E89. Print 2004 Sep. PMID 15378105
- [Background] Elliott MN, Zaslavsky AM, Goldstein E, Lehrman W, Hambarsoomians K, Beckett MK, Giordano L. Effects of survey mode, patient mix, and nonresponse on CAHPS hospital survey scores. Health Serv Res. 2009 Apr;44(2 Pt 1):501-18. doi: 10.1111/j.1475-6773.2008.00914.x. PMID 19317857